CLINICAL TRIAL: NCT00917007
Title: Measurement of Carboxyhemoglobin by Gas Chromatography as an Index of Hemolysis in ABO-compatible and Incompatible Healthy Term Newborn Infants.
Brief Title: Measurement of Carboxyhemoglobin by Gas Chromatography as an Index of Hemolysis
Status: Withdrawn | Type: Observational
Why Stopped: PI no longer at institution
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: New York State Department of Health (Other Government); Laboratory Alliance of Central New York (Unknown); Stanford University (Other)
Responsible Party: Richard H. Sills, MD, SUNY Upstate Medical University Dept of Pediatrics
Other Study IDs: IRBPHS #5803
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: ABO Incompatibility; Hemolytic Disease of Newborn; Neonatal Jaundice; Neonatal Hyperbilirubinemia
Keywords: ABO incompatibility; hemolysis; jaundice; hyperbilirubinemia; newborn
MeSH Terms: conditions — Erythroblastosis, Fetal; Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Hemolysis; Jaundice; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ABO compatible
- ABO incompatible, antiglobulin positive
- ABO incompatible, antiglobulin negative

SUMMARY:
The purpose of this research study is to more accurately measure the amount of true red blood cell breakdown (hemolysis) in newborn babies with potentially problematic blood type mismatch with their mothers (ABO incompatibility), and to examine how the true level of red blood cell destruction relates to other laboratory tests obtained in newborns with jaundice.

A better understanding of the true amount of red blood cell destruction that is caused by blood type mismatch, as well as how it relates with other laboratory tests ordered for ABO incompatibility and red blood cell destruction, would help avoid unnecessary testing, treatment and prolonged hospital stays in such babies.

DETAILED DESCRIPTION:
Clinically severe jaundice due to ABO incompatibility can occur when infants with blood type A or B are born to mothers with type O blood. An estimated 20 percent of pregnancies are ABO incompatible, but only a very small proportion of blood type A or B babies born to O type mothers develop overt ABO hemolytic disease. Despite the relative rarity of ABO hemolytic disease, it is common practice among pediatricians and family practice physicians to perform routine blood typing and antibody screening on all newborns born to type O mothers.

A very accurate and reliable laboratory measure of red blood cell destruction is the plasma carboxyhemoglobin level (COHb). COHb levels can be determined using a minute amount of blood, obtained at the same time the newborn's heel is pierced to obtain blood for the mandatory newborn screen (performed on all newborns prior to discharge) in order to avoid an additional invasive procedure.

Our hope is to determine whether routine blood typing and anti-globulin testing of infants born to type O mothers is necessary, or if these tests should instead be obtained only in the context of significant visible jaundice. This would help clarify the proper management of a very common problem in the newborn, and minimize the potential for subjecting infants of type O mothers to unnecessary blood tests, unwarranted treatment, and prolonged hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* mother blood type O
* mother Rh +
* healthy infants
* ≥37 wks gestation
* ≥ 2500 gm birth weight
* Apgar ≥5 at 1 and 5 minutes

Exclusion Criteria:

* major anomalies
* infants evaluated for sepsis or infants with transitional respiratory problems requiring >6 hrs observation in the NICU
* significant birth trauma with continued bruising and/or sequestration of blood still evident at the time of discharge
* known perinatal blood loss with hemodynamic consequences such as persistent tachycardia, need for fluid boluses or supplemental oxygen
* neonatal anemia with Hb<13.5g/dL
* known family history of hereditary hemolytic disease such as G6PD deficiency, hereditary spherocytosis or hereditary elliptocytosis

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: healthy term newborn infants of mothers with type O blood type
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Sills, MD, Principal Investigator — SUNY Upstate Medical Univeristy
Locations (2):
- United States (2):
  - Crouse Hospital, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York